CLINICAL TRIAL: NCT02391233
Title: Multimedia HIV/STI Prevention for Black Drug-Involved Women on Probation
Brief Title: Multimedia WORTH With Black Drug-Involved Women on Probation
Acronym: E-WORTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Fortune Society (Unknown); University of Pennsylvania (Other); State University of New York - Downstate Medical Center (Other); RTI International (Other); Duke University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Louisa Gilbert, Co-Director, Social Intervention Group, Columbia University School of Social Work, New York / Associate Professor, Columbia University School of Social Work, New York, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAN8409; 1R01DA038122-01 (NIH)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Sexually Transmitted Infections; HIV; Gonorrhea; Trichomonas; Chlamydia Trachomatis; Drug Use
Keywords: Effectiveness intervention; Cost-effectiveness intervention; HIV prevention; Sexually transmitted infections prevention; Multimedia evidence-based intervention; Drug-users; Black/African-American women; Probation; HIV testing
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Trichomonas Infections; Drug Misuse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV/STI Risk Reduction (Experimental): This intervention tests the comparative effectiveness of E-WORTH, streamlined HIV Testing and a 5-week multimedia intervention on primary outcomes of decreasing biologically confirmed STIs and the number and proportion of unprotected sexual acts among Black Drug-involved women on probation.
  Interventions: Behavioral: E-WORTH; Behavioral: Streamlined HIV Testing
- Streamlined HIV Testing Alone (Active Comparator): This intervention tests the comparative effectiveness of streamlined HIV Testing alone on primary outcomes of decreasing biologically confirmed STIs and the number and proportion of unprotected sexual acts among Black Drug-involved women on probation.
  Interventions: Behavioral: Streamlined HIV Testing

INTERVENTIONS:
Behavioral: E-WORTH — E-WORTH (Empowering African-American Women on the Road to Health) consists of 1 Streamlined HIV Testing session followed by 5 one-and-a-half hour group sessions that will be delivered by a probation provider at the probation site. The main multimedia components used in the E-WORTH: (1) Narrativity; (2) Skill acquisition using simulated video vignettes that provides instruction and demonstration of core skills (e.g., safer sex negotiation and problem-solving skills, technical condom use skills) using culturally congruent role models; (3) Individual interactive exercises and logs that are designed to enhance participant's recall of core knowledge and tracking of their individual progress in reducing risky behaviors and achieving risk reduction goals; and a (4) Facilitator interactive guide.
  Arms: HIV/STI Risk Reduction
Behavioral: Streamlined HIV Testing — In this intervention Black Women on Probation receive streamlined HIV Testing alone to test primary outcomes of decreasing biologically confirmed STIs and the number and proportion of unprotected sexual acts among Black Drug-involved women on probation.

SUMMARY:
The proposed study is a randomized controlled trial (RCT) that will rigorously evaluate the effectiveness and cost-effectiveness of delivering a multimedia evidence-based intervention (WORTH) and streamlined HIV testing to prevent human immunodeficiency virus (HIV) and other sexually transmitted infections (STIs) with Black/African-American (hereafter referred to as Black) women drug users in probation sites in New York City (NYC), compared to streamlined HIV testing alone. Repeated assessments will occur at baseline and 3, 6, and 12-months post intervention. The primary outcomes will be to reduce cumulative incidence of biologically confirmed STIs (i.e., Chlamydia, gonorrhea and trichomonas and the number of unprotected sex acts.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted with 420 drug-involved Black women at 5 probation sites located in communities in NYC heavily affected by HIV and STIs. Eligible women will be randomly assigned to: (1) WORTH consisting of an individual evidence-based Streamlined HIV Testing session followed by a 4-session group-based multimedia HIV intervention (WORTH) or (2) an individual Streamlined HIV Testing session alone (Streamlined HIV Testing), which will serve as the comparison condition. Both conditions will be delivered by Fortune providers at the 5 sites. Self-reported data on behavioral outcomes will be collected from participants via audio computer-assisted self-interview (ACASI). Primary STI outcomes will be measured via biological assay for infection by Neisseria gonorrhea, trichomonas, and Chlamydia trachomatis, the most common STIs found among women in NYC. Women who meet eligibility criteria will undergo a pre-intervention assessment. This assessment will last approximately 60 minutes, consisting of demographic information, history of criminal justice involvement, drug and alcohol use and dependence, sexual and drug-related HIV behaviors, HIV treatment and care, intimate partner violence, depression and posttraumatic Stress Disorder (PTSD) , service utilization, and social support. Research assistants (RAs) will schedule repeated assessments with participants that will take place at baseline and at 3, 6, and 12 months post-intervention. Each participant will be asked to obtain one vaginal specimen for STI testing by inserting a sterile Dacron-tipped swab about 2.5 inches or as far as comfortable into the vagina, rotating it for 15 to 30 seconds, and removing it. The vaginal swabs are placed into separate specimen transport packaging.

ELIGIBILITY:
Inclusion Criteria:

* She is 18 or older.
* She is currently supervised by a criminal justice entity, such as a community court or probation.
* She reports engaging in unprotected vaginal or anal sex with a male partner in the past 90 days
* She reports any illicit drug use or binge drinking in the past 6 months

Exclusion Criteria:

* Ability to speak and understand English is not sufficient to participate in assessments or intervention sessions.
* The woman's sexual activity is limited to a monogamous relationship lasting more than 12 months, and she has not engaged in any of the additional HIV risk behaviors in the past 90 days:

  * Having sex with more than one partner
  * Having sex with a partner known or suspected to be HIV positive or an injection drug user (IDU)
  * Sharing injection drug use needles or equipment
* The woman is actively trying to get pregnant/have a baby.
* Inability to complete informed consent process due to a psychiatric or cognitive impairment.
* The participant was born male.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in cumulative incidence of biologically confirmed STIs (i.e., Chlamydia, gonorrhea and trichomonas. | Baseline and 12 months post-intervention
Change in the number of unprotected sex acts | Baseline and 12 months post-intervention

SECONDARY OUTCOMES:
Change in cumulative incidence of biologically confirmed STIs (i.e., Chlamydia, gonorrhea and trichomonas as moderated by participant race, age and other socio-demographics and psychosocial client characteristics | 12-months
Change in the number of unprotected sex acts as moderated by participant race, age and other socio-demographics and psychosocial client characteristics infection rates, drug use and projected number of HIV cases averted at the 12-month follow-up. | 12-month
Comparative change in cumulative incidence of biologically confirmed STIs (i.e., Chlamydia, gonorrhea and trichomonas. | 12-month
Comparative change in the number of unprotected sex acts | 12-month
Change in cumulative incidence of biologically confirmed STIs as moderated by sociodemographics and professional training, attitudes, and self-efficacy of probation officers, administrators, and probation providers from Fortune Society | 6-month
Change in the number of unprotected sex acts as moderated by sociodemographics and professional training, attitudes, and self-efficacy of probation officers, administrators, and probation providers from Fortune Society | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Gilbert, Ph.D., Principal Investigator — Columbia University; Nabila El-Bassel, Ph.D., Principal Investigator — Columbia University; Elwin Wu, Ph.D., Study Director — Columbia University; Timothy Hunt, LCSW, Study Director — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goddard-Eckrich D, McCrimmon T, Bond K, Chang M, Hunt T, Hall J, Russo M, Ramesh V, Johnson KA, Downey DL, Wu E, El-Bassel N, Gilbert L. Effectiveness of a culturally tailored HIV intervention in promoting PrEP among black women who use drugs in community supervision programs in New York City: a randomized clinical trial. Addict Sci Clin Pract. 2024 Jul 23;19(1):55. doi: 10.1186/s13722-024-00488-0. PMID 39039560
- [Derived] Gilbert L, Goddard-Eckrich D, Chang M, Hunt T, Wu E, Johnson K, Richards S, Goodwin S, Tibbetts R, Metsch LR, El-Bassel N. Effectiveness of a Culturally Tailored HIV and Sexually Transmitted Infection Prevention Intervention for Black Women in Community Supervision Programs: A Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e215226. doi: 10.1001/jamanetworkopen.2021.5226. PMID 33835175
- [Derived] Johnson K, Gilbert L, Hunt T, Wu E, Metsch L, Goddard-Eckrich D, Richards S, Tibbetts R, Rowe JC, Wainberg ML, El-Bassel N. The effectiveness of a group-based computerized HIV/STI prevention intervention for black women who use drugs in the criminal justice system: study protocol for E-WORTH (Empowering African-American Women on the Road to Health), a Hybrid Type 1 randomized controlled trial. Trials. 2018 Sep 10;19(1):486. doi: 10.1186/s13063-018-2792-3. PMID 30201039